CLINICAL TRIAL: NCT06739798
Title: Comparison of Binocular Spectacle Prescription Versus Patching Therapy in Refractive Amblyopia Patients
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Superior University (Other)
Responsible Party: Principal Investigator, Muhammad Naveed Babur, Principal Investigator, Superior University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: MSRSW/Batch-Fall22/755
Record Dates: First submitted 2024-12-13; First posted 2024-12-18 (Actual); Last update posted 2024-12-18 (Actual); Status verified 2024-12

CONDITIONS: Amblyopia
MeSH Terms: conditions — Amblyopia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exp Group (Experimental)
  Interventions: Diagnostic Test: Exp Group
- Control Group (Active Comparator)
  Interventions: Diagnostic Test: Control Group

INTERVENTIONS:
Diagnostic Test: Exp Group — Binocular Spectacle prescription are therapeutic tools used to correct refractive errors in visually impaired patients. They improve Visual acuity as well as other visual functions in Amblyopic and visual impairment patients. They stimulate weaker eye to generate visual impulse and stimulate visual cortex to improve stereopsis and fusion.
  Arms: Exp Group
Diagnostic Test: Control Group — Patching therapy is a gold standard tool used world wide to correct visual acuity in amblyopic patients. This tool is used by occluding stronger eye with a patch or bandage or fogging lens and stimulating amblyopic eye to generate visual stimulus to motivate visual cortex.
  Arms: Control Group

SUMMARY:
This study will examine on Refractive Amblyopia patients, whose amblyopia started due to longstanding uncorrected refractive errors.

DETAILED DESCRIPTION:
There will be a comparison of two treatment methods i.e. Patching and Binocular Spectacle Prescription used to cure amblyopia patients. In binocular spectacle correction, we will slightly blur the good eye and fully correct the amblyopic eye so that binocular functions stimulate and improve after the treatment. Literature suggests that Patching improve monocular functions but there is no significant improvement in binocular functions.

ELIGIBILITY:
Inclusion Criteria:

* Anisometropic amblyopia
* Anisometropia > 1.00 D( difference between eyes in SE)
* Astigmatism >1.50 D
* VA in amblyopic eye 20/40 -20/200(6/12-6/60) or less than 20/200
* VA in the better eye or fellow eye 20/30 (6/9) or better

Exclusion Criteria:

* Strabismic amblyopia
* Deprivation amblyopia
* Isoametropic amblyopia
* History of ocular trauma, IOL implant
* Media opacity
* Any ocular/retinal pathology
* Optic nerve pathology
* Ptosis
* Any gaze control abnormalities

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 32 (Actual)
Dates: Start 2024-04-01 (Actual); Primary Completion 2024-09-01 (Actual); Study Completion 2025-03-30 (Estimated)

PRIMARY OUTCOMES:
Binocular single vision | 12 Months
  it will be measured by Worth 4 Dot test in which patient will see four lights ( two green, one red and one white light) with red and green glasses and both eyes will see at once.
  stereopsis: it will be measured grossly by seeing the fly picture at the card and fine stereopsis will be measured by different pictures available on the card. it will be assessed by wearing polarising glasses during test and see the 3D pictures."
Visual Acuity | 12 months
  it will be assessed monocularly by logMAR visual acuity chart at 4 meter distance.

CONTACTS AND LOCATIONS:
Locations (1):
- LRBT primary eyecare centre 18 Hazari, Jhang, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No